CLINICAL TRIAL: NCT00554359
Title: A Phase I, Randomized, Double-Blind, Dose Escalation Trial of the Safety and Pharmacokinetics of a Single Intravenous Injection of I5NP in Patients Undergoing Major Cardiovascular Surgery
Brief Title: A Dose Escalation and Safety Study of I5NP in Patients Undergoing Major Cardiovascular Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Mike Johnston, Director of Regulatory Affairs, Quark Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QRK.002
Record Dates: First submitted 2007-11-04; First posted 2007-11-06 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Injury of Kidney; Acute Renal Failure
Keywords: Acute Kidney Injury; Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I5NP drug (Experimental)
  Interventions: Drug: I5NP (a small interfering RNA)
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: I5NP (a small interfering RNA) — Single IV injection of experimental drug
  Arms: I5NP drug
Drug: placebo — Single IV injection of saline
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, dose escalation, safety and pharmacokinetic study. The study will be conducted in approximately 8-10 centers in the United States and Switzerland. Up to 32 patients who have undergone major cardiovascular surgery will participate. Patients will receive a single IV injection of I5NP or placebo following cardiovascular surgery. I5NP will be administered 4 hours (+/- 30 minutes) following removal of the cardiopulmonary bypass machine (CBM).

The duration of the study is approximately 44 days, inclusive of a 14 day screening period. Patients will be contacted by phone at 6 and 12 months for follow-up questions. Patient visits are screening, day of surgery, hospital in-patient Days 1, 2, 3 and Day 7 or hospital discharge. Safety follow-up will continue until 30 days post-surgery. 2 phone calls will be made at 6 and 12 months after date of surgery.

DETAILED DESCRIPTION:
The drug (I5NP) is a small interfering RNA that is being developed to protect patients from acute kidney injury after cardiac bypass surgery. This first-in-man study will test the safety of I5NP and measure how long the drug stays in the blood stream after injection. This study is not meant to test if I5NP protects kidneys from the damage that may occur in rare cases during surgery. Another purpose of this dose escalation study is to find out the right dose of the experimental drug to be given to study subjects in future studies. Even though there were no harmful effects seen in the animals tested, we do not know what side effects the experimental drug might cause in humans.

ELIGIBILITY:
Inclusion Criteria (before surgery):

* Patient age between 21 years and 85 years old
* Patient is capable of giving consent
* Patient is willing and able to comply with the visit schedule and study procedures including post-hospitalization discharge follow-up
* Patient is undergoing non-emergent coronary artery bypass graft (CABG) and/or valve replacement surgery
* Patient has a cumulative score of 0 to 8 on the Cleveland Clinic Foundation (CCF) Acute Kidney Injury (AKI) risk factor scale
* The patient reports that they are up to date and have had normal findings on their age- and sex-appropriate cancer screening, per American Cancer Society guidelines, for breast cancer, cervical cancer, rectal cancer, and prostate cancer. If a patient is not up to date, the relevant screening test must be performed and a normal result documented prior to dosing.

Inclusion Criteria (during surgery):

* Patient must have been on cardiopulmonary bypass machine (CBM)

Inclusion Criteria (after surgery):

* Patient must be in the ICU for dosing to facilitate study procedures including PK blood draws and PK urine sampling

Exclusion Criteria (before surgery):

* Patient has undergone any organ transplant
* Patient who has had cancer or may be predisposed to develop cancers such as those with family history of cancers in multiple relatives {i.e., Familial Polyposis Coli, those with family history of Von Hippel Landau disease (associated with renal cell cancers and renal cysts) and those with family history of Li-Fraumeni syndrome (associated with inherited mutations of the p53 tumor-suppressor gene)}
* Patient has a history of any abnormality on chest X-ray that could represent a malignancy
* Patient has a clinically significantly elevated pancreatic and/or hepatic enzyme level, defined as any grade 2, 3 or 4 value according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 3.0
* Patient has an underlying medical condition which increases the risk of perioperative complications, such as poorly controlled diabetes mellitus or hypertension or significant chronic obstructive pulmonary disease (COPD)
* Women of childbearing potential are to be excluded from this study. Every female subject is considered of childbearing potential unless she has had sterilization surgery, or is post-menopausal.

  * Women 21-59, post-menopausal is defined as no menses for at least 12 months and an elevated follicle stimulating hormone (FSH) level.
  * Women 60-85, post-menopausal is defined as no menses in at least 12 months.
* Patient has participated in a study of an experimental therapy in the last 30 days
* Patient is currently receiving immunosuppressive therapy [this criterion does NOT apply to topical steroids and inhalation steroids for chronic obstructive pulmonary disease (COPD) and/or asthma]
* Patient requires pre-operative dialysis or is currently on dialysis
* Patient is undergoing aortic aneurism repair
* Pre-operative extracorporeal membrane oxygenation
* Pre-operative tracheotomy, or mechanical ventilation
* Patient has Intra-Arterial Balloon Pump (IABP) or other Left Ventricular Assist Device (LVAD)
* Evidence that patient is experiencing possible AKI prior to surgery, defined as a > 1.5 times increase in serum creatinine from screening to any time prior to surgery
* Baseline serum creatinine > 3.0 mg/dL and/or an estimated GFR of < 30 mL/min/1.73 m2, as calculated by the Modification of Diet in Renal Disease [MDRD] Study equation: eGFR (mL/min/1.73 m2) = [186 x (SCr)] - [1.154 x (Age)] - [0.203 x (0.742 if female or 1.210 if African-American female)] where SCr: serum creatinine in mg/dL and age is in years
* Patient has comfort measures only or do not resuscitate (DNR) status
* Patient is participating in a concurrent interventional study
* Patient has received intravenous contrast material < 48 hours prior to surgery
* In the opinion of the investigator a pre-operative concomitant disease or clinical finding such as an abnormality in clinical lab results, chest X-ray, EKG, or physical examination finding that significantly raises the risk of perioperative complications precludes dosing of the patient

Exclusion Criteria (during surgery):

* Patient on CBM for > 3 hours
* Patient experienced major blood loss (>15 units)
* Use of balloon pump or other LVAD during surgery;
* In the opinion of the investigator, an intra-operative complication precludes dosing of the patient

Exclusion Criteria (2-3 days post-removal of CBM):

* Cardiac Index < 2.1 L/min/m2 (applies only to patients with a Swan-Ganz or other PA catheter)
* Patient has a body temperature ≥ 40 °C
* Use of IABP post-surgery
* Fluid imbalance in excess of 15 liters
* PaO2:FiO2 < 250
* Patient receiving ≥ 3 concurrent vasopressors to maintain hemodynamic stability
* In the opinion of the investigator a post-operative complication precludes dosing of the patient

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities (DLTs) observed among 4 cohorts of 4-8 patients per cohort | Reviewed at the conclusion of each cohort
Pharmacokinetics | Immediately following injection through 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Polinsky, M.D., Study Director — Quark Pharmaceuticals
Locations (11):
- United States (6):
  - George Washington University, Washington D.C., District of Columbia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Switzerland (2):
  - University Hospital of Geneva, Geneva
  - Lausanne University Hospital (CHUV), Lausanne